CLINICAL TRIAL: NCT03321071
Title: Interventions to Promote Healthy Lifestyle and Academic Performance in Children During the Summer Months.
Brief Title: Healthy Summer Learners
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, R. Glenn Weaver, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00065094
Record Dates: First submitted 2017-08-25; First posted 2017-10-25 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-01

CONDITIONS: Overweight and Obesity; Academic Acheivement
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Summer Learners (Experimental): Similar to typical summer day camp procedures, students attending Healthy Summer Learners will be dropped-off and picked-up at camp. The physical activity component of the program was designed with the expertise and input from B&G Club youth program staff. The academic component was informed by school district personnel. The program was also designed to be analogous to typical summer day camp program in terms of operating weeks (10 weeks) length of program day (i.e., 8am-5pm), and program component time blocks (~45min-1hr time blocks).
  Interventions: Behavioral: Healthy Summer Learners
- 21st Century Learning Center (Active Comparator): Children in this condition will attend a 21st Century Summer Learning Program.
  Interventions: Behavioral: 21st Century Summer Learning Center
- Passive control (No Intervention): Children in this condition will not attend a summer program.

INTERVENTIONS:
Behavioral: Healthy Summer Learners — Physical Activity Component. The physical activity component of Healthy Summer Learners is designed to engage children in moderate-to-vigorous physical activity (MVPA) for at least 50% of the time. With 3 hours each day dedicated to physical activity, this translates into children accumulating 90 minutes of MVPA daily. This is 30 minutes above the 60 minutes of MVPA each day recommended by the Physical Activity Guidelines for Americans.
  Nutrition Component. The nutrition component of Healthy Summer Learners is designed to provide healthy snacks and meals and nutrition education via standardized pre-existing curricula.
  Food/Beverage Guidelines. Meals will follow the USDA Nutrition Standards for the National School Lunch and School Breakfast Programs.
  Academic Component. The academic component will consist of existing, effective academic programs focused on Math and Reading.
  Arms: Healthy Summer Learners
Behavioral: 21st Century Summer Learning Center — Children in this condition will attend a 21st Century Summer Learning Program.
  Arms: 21st Century Learning Center

SUMMARY:
Summer vacation represents a "window of vulnerability" where dramatic declines in both health and academics occur for elementary age children. Currently, there are no summer programs that incorporate curriculum addressing both unhealthy weight gains and academic achievement simultaneously. This work represents an important step towards addressing important public health goals - obesity and learning - through a comprehensive program delivered during a timeframe - summer vacation - where substantial and long-lasting negative effects occur.

DETAILED DESCRIPTION:
Summer vacation represents an important time away from the school setting for a majority of children attending public school in the US. This break is characterized by large amounts of free time and involvement in a wide variety of formal and informal activities, time spent with friends and family, and travel. Yet for many children, particularly those from low-income households, summer vacation represents a "window of vulnerability" in which dramatic declines in both health and academics occur. During the summer months (typically 3 months) children gain a larger amount of body weight compared to the amount of weight gained over the school year, and weight gain during summer reverses weight losses achieved during school. For academics, it is well established that children from low-income households experience greater declines in reading and math during the summer than their middle-to-upper income peers. Numerous programs that address these issues currently exist (e.g., summer school, summer weight loss or fitness programs). However, these programs are designed and delivered at the expense of the promotion or prevention of the other - academic focus without health or health focus without academics. Our long-term goal is to develop summer programming for widespread dissemination that addresses both lifestyle behaviors (i.e., physical activity and nutrition) and academic performance. The objective of the proposed study is to establish the effectiveness of an innovative "Healthy Summer Learners" (HSL) program for low-income, minority children. The rationale for the proposed research is that no summer programs incorporate curriculum that addresses both unhealthy weight gains and academic achievement simultaneously. This study seeks to fill this void by testing a prototype learning and health-oriented summer program focused on promoting physical activity and nutrition, along with content that provides quality learning experiences to develop reading and math skills. To accomplish this objective, this study will evaluate over 2 summers the effectiveness of a 6-week Healthy Summer Learners program delivered within a Boys & Girls Club summer camp using a randomized design in a sample of rising 2nd, 3rd, and 4th graders. The aims of the study are Aim 1: Evaluate the impact of Healthy Summer Learners on children's weight gain and academic performance from beginning (end of Spring school year) to the end of summer (beginning of Fall school year), and Aim 2: Evaluate the feasibility and acceptability of Healthy Summer Learners to children, parents, and program staff.

ELIGIBILITY:
Inclusion Criteria:

* MAP scores are norm referenced based on typical grade level scores. Students that have scored between the 25th and 75th percentile will be eligible to participate in the study.

Exclusion Criteria:

* children with severe intellectual or physical disabilities

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We will not share IPD data.

REFERENCES:
- [Derived] von Klinggraeff L, Dugger R, Brazendale K, Hunt ET, Moore JB, Turner-McGrievy G, Vogler K, Beets MW, Armstrong B, Weaver RG. Healthy Summer Learners: An explanatory mixed methods study and process evaluation. Eval Program Plann. 2022 Jun;92:102070. doi: 10.1016/j.evalprogplan.2022.102070. Epub 2022 Mar 17. PMID 35339766
- [Derived] Dugger R, Brazendale K, Hunt ET, Moore JB, Turner-McGrievy G, Vogler K, Beets MW, Armstrong B, Weaver RG. The impact of summer programming on the obesogenic behaviors of children: behavioral outcomes from a quasi-experimental pilot trial. Pilot Feasibility Stud. 2020 May 28;6:78. doi: 10.1186/s40814-020-00617-x. eCollection 2020. PMID 32514369

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Summer Learners: Similar to typical summer day camp procedures, students attending Healthy Summer Learners will be dropped-off and picked-up at camp. The physical activity component of the program was designed with the expertise and input from B&G Club youth program staff. The academic component was informed by school district personnel. The program was also designed to be analogous to typical summer day camp program in terms of operating weeks (6 weeks) length of program day (i.e., 8am-5pm), and program component time blocks (~45min-1hr time blocks).
  Healthy Summer Learners: Physical Activity Component. The physical activity component of Healthy Summer Learners is designed to engage children in moderate-to-vigorous physical activity (MVPA) for at least 50% of the time. With 3 hours each day dedicated to physical activity, this translates into children accumulating 90 minutes of MVPA daily. This is 30 minutes above the 60 minutes of MVPA each day recommended by the Physical Activity Guidelines for Americans.
  Nutrition Component. The nutrition component of Healthy Summer Learners is designed to provide healthy snacks and meals and nutrition education via standardized pre-existing curricula.
  Food/Beverage Guidelines. Meals will follow the USDA Nutrition Standards for the National School Lunch and School Breakfast Programs.
  Academic Component. The academic component will consist of existing, effective academic programs focused on Math and Reading.
- 21st Century Learning Center: The 21C is a federally funded program providing academic enrichment opportunities for students who attend low-performing schools. Students enrolled in 21C will attend the same school as children enrolled in HSL. The 21C will operate daily (Monday-Thursday) from 8:30-14:00 for four weeks during the summer. The program day will consist of academic sessions in the morning and afternoon (9:00-11:30 & 12:30-13:45) and one hour of physical activity before lunch (11:30-12:30). All participants will be provided a USDA Summer Feeding Program compliant breakfast (8:30-9:00) and lunch (11:30-12:30).
- Passive Control: Children in this condition will not attend a summer program but will be followed from baseline to followup (i.e., 12 weeks)
Period: Overall Study
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Started | 60 | 60 | 60
Completed | 57 | 51 | 55
Not Completed | 3 | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Healthy Summer Learners: Similar to typical summer day camp procedures, students attending Healthy Summer Learners will be dropped-off and picked-up at camp. The physical activity component of the program was designed with the expertise and input from B&G Club youth program staff. The academic component was informed by school district personnel. The program was also designed to be analogous to typical summer day camp program in terms of operating weeks (10 weeks) length of program day (i.e., 8am-5pm), and program component time blocks (~45min-1hr time blocks).
  Healthy Summer Learners: Physical Activity Component. The physical activity component of Healthy Summer Learners is designed to engage children in moderate-to-vigorous physical activity (MVPA) for at least 50% of the time. With 3 hours each day dedicated to physical activity, this translates into children accumulating 90 minutes of MVPA daily. This is 30 minutes above the 60 minutes of MVPA each day recommended by the Physical Activity Guidelines for Americans.
  Nutrition Component. The nutrition component of Healthy Summer Learners is designed to provide healthy snacks and meals and nutrition education via standardized pre-existing curricula.
  Food/Beverage Guidelines. Meals will follow the USDA Nutrition Standards for the National School Lunch and School Breakfast Programs.
  Academic Component. The academic component will consist of existing, effective academic programs focused on Math and Reading.
- Total: Total of all reporting groups
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 60 | 60 | 180
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (1.0) | 7.9 (1.0) | 8.0 (1.0) | 7.9 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 43 | 33 | 107
  Male | 29 | 17 | 27 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 55 | 56 | 56 | 167
  White | 5 | 4 | 4 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 60 | 180
BMI z-score [Mean (Standard Deviation); unit: units on a scale] — Centers for Disease Control age and sex-specific Body Mass Index z-scores A z-score of 0 represents the population mean Higher or lower z-scores could represent better or worse outcomes as too low could be underweight and too high could indicate overweight or obesity.
  Children above the 85th percentile are considered overweight while children above the 95th percentile are considered obese
  units on a scale | 0.99 (1.1) | 0.99 (1.1) | 0.95 (1.1) | 0.98 (1.1)
Measures of Academic Progress Reading Scores [Mean (Standard Deviation); unit: units on a scale] — Created by the Northwest Evaluation Association (www.nwea.org), MAP results are widely accepted and used extensively in school-aged children. Scores are reported using the Rasch Unit Scale, a curriculum scale developed using Item Response Theory that estimates student achievement. The Rasch Unit Scale ranges from 140-300 and are norm referenced based on grade. Higher scores indicate better reading profeciency.
  units on a scale | 190.8 (12.0) | 192.6 (13.5) | 194 (11.6) | 192.5 (12.4)
PACER Laps Completed [Mean (Standard Deviation); unit: Laps] — For the PACER test children were instructed to run from one cone marker to another cone placed at a length of 20 meters. Music and voice instructions were used to prompt children to run and stop within an allotted amount of time. As the test progressed, the allotted time to run the 20 meters incrementally decreased. If the child failed to reach the cone/marker within the allotted time frame on two occasions the test was ended, and the laps score was recorded. More completed laps indicates higher cardiorespiratory fitness.
  Laps | 13.5 (7.4) | 13.5 (7.4) | 11.6 (6.9) | 12.9 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index (BMI) Z-score
Description: Measure Description: Centers for Disease Control age and sex-specific Body Mass Index z-scores. A z-score of 0 represents the population mean. Higher or lower z-scores could represent better or worse outcomes as too low could be underweight and too high could indicate overweight or obesity.
  Children above the 85th percentile are considered overweight while children above the 95th percentile are considered obese
Time Frame: Body mass index will be collected in the spring academic semester up to 6 weeks prior to attending HSL and the fall academic semester up to 6 weeks after attending HSL
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 60
z-score | 0.03 [-0.03 to 0.09] | 0.02 [-0.03 to 0.08] | 0.06 [0.01 to 0.12]

2. Primary Outcome: Change in Measures of Academic Progress Reading Scores
Description: Measure Description: Created by the Northwest Evaluation Association (www.nwea.org), MAP results are widely accepted and used extensively in school-aged children. Scores are reported using the Rasch Unit Scale, a curriculum scale developed using Item Response Theory that estimates student achievement. The Rasch Unit Scale ranges from 140-300 and are norm referenced based on grade. Higher scores indicate better reading profeciency.
Time Frame: MAP reading scores will be collected in the spring academic semester up to 6 weeks prior to attending HSL and the fall academic semester up to 6 weeks after attending HSL
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 1.8 [-0.5 to 4.2] | 0.7 [-1.5 to 2.8] | 0.9 [-1.4 to 3.2]

3. Secondary Outcome: Average Minutes Per Day Spent in Moderate to Vigorous Physical Activity During the Summer on Days Attending a Program and Not Attending a Program
Description: Moderate to vigorous physical activity will be collected via a wrist placed Fitbit. Negative numbers mean the behavior decreased on days attending while positive numbers indicate the behavior increased on days attending. No change is indicated for the passive control as they did not attend a program. Passive control never attended a structured summer program thus no change can be calculated.
Time Frame: Moderate to vigorous physical activity will be collected daily from baseline to 12 weeks
Population: data not collected for the passive control arm because they did not attend a structured summer program
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 0
minutes per day | 51.2 [33.3 to 69.0] | 15.0 [6.6 to 23.4] |

4. Secondary Outcome: Average Minutes Per Day Spent in Sedentary Behavior During the Summer on Days Attending a Program and Not Attending a Program
Description: Sedentary time will be collected via a wrist placed Fitbit. Negative numbers mean the behavior decreased on days attending while positive numbers indicate the behavior increased on days attending. No change is indicated for the passive control as they did not attend a program. Passive control never attended a structured summer program thus no change can be calculated.
Time Frame: Sedentary time will be collected daily from baseline to 12 weeks
Population: data not collected for the passive control arm because they did not attend a structured summer program
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 0
minutes per day | -138.8 [-171.7 to -105.9] | -80.2 [-112.3 to -48.2] |

5. Secondary Outcome: Average Minutes Per Day Screen Time During the Summer on Days Attending a Program and Not Attending a Program
Description: Screen time will be collected via parent proxy report during the summer. Passive control never attended a structured summer program thus no change can be calculated.
Time Frame: Screen time will be collected twice weekly from baseline to 12 weeks
Population: data not collected for the passive control arm because they did not attend a structured summer program
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 0
minutes per day | -44.0 [-78.6 to -9.4] | -57.3 [-92.0 to -22.6] |

6. Secondary Outcome: Average Number of Healthy Foods Consumed/Day on Days Attending a Program and Not Attending a Program
Description: Diet will be collected via food frequency questionnaires and the number of healthy and unhealthy foods consumed will be calculated. Negative numbers mean the number of healthy foods consumed decreased on days attending while positive numbers indicate the number of healthy foods consumed increased on days attending. No change is indicated for the passive control as they did not attend a program. Passive control never attended a structured summer program thus no change can be calculated.
Time Frame: Diet will be collected twice weekly from baseline to 12 weeks
Population: data not collected for the passive control arm because they did not attend a structured summer program
Measure: Mean (95% Confidence Interval); unit: number of health foods consumed per day
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 0
number of health foods consumed per day | 0.06 [-0.19 to 0.32] | -0.17 [-0.46 to 0.11] |

7. Secondary Outcome: Average Minutes Per Day of Sleep During the Summer on Days Attending a Program and Not Attending a Program
Description: Sleep time will be collected via a wrist placed Fitbit. Negative numbers mean the behavior decreased on days attending while positive numbers indicate the behavior increased on days attending. No change is indicated for the passive control as they did not attend a program.
Time Frame: Sleep will be collected daily from baseline to 12 weeks
Population: data not collected for the passive control arm because they did not attend a structured summer program
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 0
minutes per day | -20.6 [-43.9 to 2.7] | -16.2 [-31.5 to -0.9] |

8. Secondary Outcome: Average Minutes Per Day Shift in Sleep Onset During the Summer on Days Attending a Program and Not Attending a Program.
Description: Sleep onset will be collected via a wrist placed Fitbit. Negative numbers indicate sleep onset was earlier on days attending while positive numbers indicate sleep onset was later on days attending. No change is indicated for the passive control as they did not attend a program.
Time Frame: Sleep onset will be collected daily from baseline to 12 weeks
Population: data not collected for the passive control arm because they did not attend a structured summer program
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 0
minutes per day | -52.9 [-81.9 to -24.0] | -88.2 [-115.0 to -61.3] |

9. Secondary Outcome: Average Minutes Per Day Shift in Sleep Offset During the Summer on Days Attending a Program and Not Attending a Program
Description: Sleep offset will be collected via a wrist-placed Fitbit. Negative numbers mean sleep offset was earlier on days attending while positive numbers indicate sleep offset was later on days attending. No change is indicated for the passive control as they did not attend a program.
Time Frame: Sleep offset will be collected daily from baseline to 12 weeks
Population: data not collected for the passive control arm because they did not attend a structured summer program
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 0
minutes per day | -95.5 [-122.6 to -68.3] | -104.8 [-124.8 to -84.8] |

10. Secondary Outcome: Average Minutes Per Day Shift in Sleep Midpoint During the Summer on Days Attending a Program and Not Attending a Program
Description: Sleep midpoint will be collected via a wrist placed Fitbit. Negative numbers mean midpoint was earlier on days attending while positive numbers indicate midpoint was later on days attending. No change is indicated for the passive control as they did not attend a program.
Time Frame: Sleep midpoint will be collected daily from baseline to 12 weeks
Population: data not collected for the passive control arm because they did not attend a structured summer program
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 0
minutes per day | -73.3 [-102.4 to -44.3] | -99.5 [-148.2 to -50.7] |

11. Other Pre Specified Outcome: Change in Progressive Aerobic Cardiovascular Endurance Run Laps
Description: Children were instructed to run from one cone marker to another cone placed at a length of 20 meters. Music and voice instructions were used to prompt children to run and stop within an allotted amount of time. As the test progressed, the allotted time to run the 20 meters incrementally decreased. If the child failed to reach the cone/marker within the allotted time frame on two occasions the test was ended, and the laps score was recorded.
Time Frame: Change in Progressive Aerobic Cardiovascular Endurance Run Laps will be collected in the spring academic semester up to 6 weeks prior to attending HSL and the fall academic semester up to 6 weeks after attending HSL
Measure: Least Squares Mean (95% Confidence Interval); unit: Laps
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
Number analyzed (Participants) | 60 | 60 | 60
Laps | -0.1 [-1.8 to 1.5] | 1.3 [0.3 to 2.9] | -0.1 [-1.7 to 1.5]

ADVERSE EVENTS:
Time Frame: Data were collected for the 12 weeks that each participant was enrolled in the project (baseline to follow-up).
Description: The participants were healthy children
Arm/Group | Healthy Summer Learners | 21st Century Learning Center | Passive Control
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT03321071/Prot_SAP_000.pdf